CLINICAL TRIAL: NCT02894268
Title: Doxycycline- and Furazolidone-containing Quadruple Regimen is Superior of Tailored Therapy as Rescue Treatment for Helicobacter Pylori Infection After Failure of Several Therapy
Brief Title: Doxycycline- and Furazolidone-containing Quadruple Regimen is Superior of Tailored Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Weiling Hu, MD,PhD, Clinical Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160513-1
Record Dates: First submitted 2016-08-25; First posted 2016-09-09 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Doxycycline; Furazolidone; Esomeprazole; bismuth tripotassium dicitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (Experimental): esomeprazole (E) 20 mg, doxycycline (D) 100mg, furazolidone (F) 100 mg, and colloidal bismuth subcitrate (B) 100 mg
  Interventions: Drug: Doxycycline; Drug: Furazolidone; Drug: Esomeprazole; Drug: Colloidal Bismuth Subcitrate
- Regimen B (Active Comparator): two sensitivity antibiotics based on antibiotic sensitivity of helicobacter pylori culture, colloidal bismuth subcitrate (B) 100 mg, esomeprazole (E) 20 mg
  Interventions: Drug: Esomeprazole; Drug: Colloidal Bismuth Subcitrate; Drug: Sensitivity antibiotics

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100g po bid
  Other Names: Vibramycin
  Arms: Regimen A
Drug: Furazolidone — Furazolidone 100mg po bid
  Other Names: Giarlan
  Arms: Regimen A
Drug: Esomeprazole — Esomeprazole 20mg po bid
  Other Names: Nexium
Drug: Colloidal Bismuth Subcitrate — Bismuth 20mg po bid
  Other Names: PIDI
Drug: Sensitivity antibiotics — Two antibiotics based on antibiotic sensitivity of H.pylori culture, including amoxicillin, clarithromycin, metronidazole, levofloxacin, tetracycline and furazolidone.
  Arms: Regimen B

SUMMARY:
Doxycycline- and Furazolidone-containing Quadruple Regimen can be a successful rescue treatment for Helicobacter pylori Infection patients after Failure of several therapy. It is superior of tailored therapy as rescue treatment for helicobacter pylori Infection after failure of several therapy.

DETAILED DESCRIPTION:
This study is a prospective, multiple centers, randomized trial. Patients who had failed in previous H. pylori eradication treatment that more than two times will be enrolled in Sir Run Run Shaw Hospital.

Pretreatment H. pylori status will be defined by a positive 13 C-urea breath test (13 C-UBT). Patients who had received bismuth compounds, acid inhibitor, or antibiotics during 4 weeks before 13 C-UBT are excluded. Other exclusion criteria included upper gastrointestinal surgery, malignancy, and evidence of blood dyscrasia.

After the patient is enrolled the patient will sign the informed consent and receive gastroscopy. More than four biopsy will be given including two in antrum and two in gastric body. One pair of biopsy sample will be sent for the pathology and the other pair is used for H.pylori culture and antibiotics sensitivity. After we get the result of antibiotics sensitivity the patient will be divided randomly into two groups, Regimen A, Regimen B.

The Regimen A includes esomeprazole (E) 20 mg, doxycycline (D) 100mg, furazolidone (F) 100 mg, and colloidal bismuth subcitrate (B) 100 mg . All drugs are taken twice a day for 14 days. The Regimen B includes two antibiotics based on antibiotic sensitivity of helicobacter pylori culture, colloidal bismuth subcitrate (B) 100 mg, esomeprazole (E) 20 mg. The esomeprazole and bismuth are taken half an hour before a meal and antibiotics after the meal.

All patients are asked to quit smoking and drinking and forbid eating foods rich in tyramine (e.g., chicken, cheese, pickles, lentils, beans) and seafood during and in 1 week after the treatment.

Patients will be followed up at the 1st day, 14th day, and 4 weeks after the treatment, respectively, and all side effects will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. A positive 13 C-urea breath test
2. Formal H.pylori treatment more than two times
3. Age >18 years

Exclusion Criteria:

1. Bismuth compounds, acid inhibitor, or antibiotics during 4 weeks before the patient is enrolled
2. Allergic to the medications
3. Upper gastrointestinal surgery history
4. Serious heart insufficiency, liver insufficiency, renal insufficiency and other serious medical problems
5. Evidence of blood dyscrasia
6. Pregnant and lactating women
7. Can't express his complain correctly and can't cooperate with the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 42 days after start of therapy
  Repeat 13-Urea breath test 42 days after H.pylori eradication

SECONDARY OUTCOMES:
Clinical response as measured by Number of participants whose symptoms disappear or improve after eradication treatment | 14 days and 42 days after H.pylori eradication
  Number of participants whose symptoms disappear or improve after eradication treatment.
Side effects | 14 days after start of therapy
  Adverse Events That Are Related to Eradication Treatment
Adherence rate | 14 days after start of therapy
  Number of patients who take at least 80% drugs

CONTACTS AND LOCATIONS:
Overall Officials: Weiling Hu, Attending, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Gao W, Cheng H, Zhang X, Hu F. Tetracycline- and furazolidone-containing quadruple regimen as rescue treatment for Helicobacter pylori infection: a single center retrospective study. Helicobacter. 2014 Oct;19(5):382-6. doi: 10.1111/hel.12143. Epub 2014 May 21. PMID 24849129
- [Result] Ciccaglione AF, Cellini L, Grossi L, Manzoli L, Marzio L. A Triple and Quadruple Therapy with Doxycycline and Bismuth for First-Line Treatment of Helicobacter pylori Infection: A Pilot Study. Helicobacter. 2015 Oct;20(5):390-6. doi: 10.1111/hel.12209. Epub 2015 Mar 20. PMID 25801708